CLINICAL TRIAL: NCT00276211
Title: Diffusionsvægtet MR Skanning Med Henblik på axillære Lymfeknudemetastaser Hos Patienter Med primær Mammacancer - et Pilotstudie
Brief Title: Diffusion Weighted MRI for Lymphnodes in the Axilla
Status: Completed | Type: Observational
Sponsor: Copenhagen University Hospital at Herlev (Other)
Responsible Party: Copenhagen University Hospital at Herlev, Region H
Other Study IDs: KA-20051023
Record Dates: First submitted 2006-01-06; First posted 2006-01-13 (Estimated); Last update posted 2009-01-28 (Estimated); Status verified 2006-01

CONDITIONS: Breast Cancer
Keywords: MRI diffusion mamma cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
This study is going to compare diffusionweigthed MRI scanning to the result of surgey in patients with metastasis from brestcancer in the axilla

ELIGIBILITY:
Inclusion Criteria:

Newly diagnosed breast cancer patients, where ultrasound and cytologi has proved one or more malignant lymphnodes in the axilla.

Exclusion Criteria:

Pacemaker metal in the body claustrphobia psychiatry patients pregnancy age below 18 years

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2006-01; Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jakob M Møller, M.Sc., Principal Investigator — Copenhagen University Hospital at Herlev
Locations (1):
- Department of Radiology, Herlev University Hospital, Herlev, Denmark